CLINICAL TRIAL: NCT01446640
Title: PhaseⅠ/ⅡTrial of Autologous Bone Marrow Derived Mesenchymal Stem Cells to Patients With Spinal Cord Injury.
Brief Title: Mesenchymal Stem Cells Transplantation to Patients With Spinal Cord Injury
Acronym: MSC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-2011-09
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2011-10-05 (Estimated); Status verified 2011-10

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSC (Experimental): Intravenous combined with intrathecal administration of autologous bone marrow derived mesenchymal stem cells to patients with spinal cord injury.
  Interventions: Biological: bone marrow derived mesenchymal stem cells

INTERVENTIONS:
Biological: bone marrow derived mesenchymal stem cells — Intravenous administration of up to 1x10^6 MSCs per kg; intrathecal administration of up to 1x10^6 MSCs per kg.
  Other Names: Mesenchymal Stem Cells; Multipotent Mesenchymal Stem Cells; Multipotent Mesenchymal Stromal Cells

SUMMARY:
The study is a phase I/II trial designed to establish the safety and efficacy of intravenous combined with intrathecal administration of autologous bone marrow derived mesenchymal stem cells to patients with spinal cord injury.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a traumatic disorder resulting in a functional deficit that usually leads to severe and permanent paralysis. Pharmacological and rehabilitation therapies to SCI get limited effect. Another promising therapeutic approaches for SCI is cellular transplantation. Cell types used in SCI therapy include Schwann cells, olfactory ensheathing cells and adult stem cells, such as neural stem cells, umbilical cord blood derived cells, mesenchymal stem cells (MSCs) or induced pluripotent stem cells. There are not yet conclusive evidences on which types of glial or adult stem cells are most effective in SCI treatment.

MSC have been shown to promote anatomical and functional recovery in animal models of SCI by promoting tissue sparing ,axonal regeneration, and remyelination. Therapeutic effects of MSCs are primarily due to the secretion of soluble factors and the provision of extracellular matrix that provide protection and support repair. MSC are attractive candidates for transplantation into human patients because they can be easily harvested, expanded and banked, or derived directly from the patient allowing for autologous transplantation, obviating the need for immune suppression.

The clinical translation of cellular transplantation strategies requires a safe and efficient means of cellular delivery. In animal models of SCI, the most common delivery is direct injection into the injury site, which allows a defined number of cells to be delivered, but risks further injuring the cord. Less invasive methods for cell delivery have been investigated, including intravascular delivery (intravenous (IV) and intra-arterial) and delivery into the cerebrospinal fluid (intrathecal). These minimally-invasive techniques decrease the risk to the patient and allow delivery of multiple cell doses. Maybe intrathecal administration is superior to IV delivery, cell engraftment and tissue sparing were significantly better after intrathecal delivery, but more researches are needed for get conclusion.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic spinal cord injury at the thoracic or lumbar level.
* Age 16 to 60.
* American Spinal Injury Association Impairment Scale A or B.
* Time between injury and enrollment greater than 2 weeks and less than 1 year.
* Patients must have organ function as defined below:

total bilirubin within normal institutional limits (NV: 0.0-20.5 umol/L); AST(SGOT)/ALT(SGPT) <2.5 × institutional upper limit of normal AST (NV: 0-35 U/L); ALT (NV: 0-40 U/L) ; Creatinine within normal institutional limits (NV: 53-106 umol/L) or Creatinine clearance >1.25 ml/s for patients with creatinine levels above institutional normal.

* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents within 4 weeks of study entry.
* History of allergic reactions attributed to compounds of similar biologic composition to mesenchymal stem cells.
* Primary hematologic diseases.
* Open injuries.
* Psychiatric, addictive or any other disorder that compromises ability to give a truly informed consent.
* Malignancy within the last 5 years.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (defined as invasive fungal infection and progressive CMV viremia), symptomatic congestive heart failure (NYH class III and IV), unstable angina pectoris, or cardiac arrhythmia.
* Pregnant or breastfeeding women.
* HIV-positive patients.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 1 month after transplantation

SECONDARY OUTCOMES:
Electromyogram and Electroneurophysiologic test | 1 month after transplantation
  somatosensory and motor evoked potentials
Muscle strength assessment | 1 month after transplantation
  Assessed by the Frankel scale.
Motor and sensory assessment | 1 month after transplantation
  Assessed by ASIA score
Electromyogram and Electroneurophysiologic test | 3 months after transplantation
  somatosensory and motor evoked potentials
Muscle strength assessment | 3 months after transplantation
  Assessed by the Frankel scale.
Motor and sensory assessment | 3 months after transplantation
  Assessed by ASIA score
Electromyogram and Electroneurophysiologic test | 6 months after transplantation
  somatosensory and motor evoked potentials
Muscle strength assessment | 6 months after transplantation
  Assessed by the Frankel scale.
Motor and sensory assessment | 6 months after transplantation
  Assessed by ASIA score
Electromyogram and Electroneurophysiologic test | 12 months after transplantation
  somatosensory and motor evoked potentials
Muscle strength assessment | 12 months after transplantation
  Assessed by the Frankel scale.
Motor and sensory assessment | 12 months after transplantation
  Assessed by ASIA score

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xiao, MD, Study Director — Guangzhou General Hospital of Guangzhou Military Command
Locations (1):
- Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Hernandez J, Torres-Espin A, Navarro X. Adult stem cell transplants for spinal cord injury repair: current state in preclinical research. Curr Stem Cell Res Ther. 2011 Sep;6(3):273-87. doi: 10.2174/157488811796575323. PMID 21476980
- [Background] Paul C, Samdani AF, Betz RR, Fischer I, Neuhuber B. Grafting of human bone marrow stromal cells into spinal cord injury: a comparison of delivery methods. Spine (Phila Pa 1976). 2009 Feb 15;34(4):328-34. doi: 10.1097/BRS.0b013e31819403ce. PMID 19182705
- [Background] Sheth RN, Manzano G, Li X, Levi AD. Transplantation of human bone marrow-derived stromal cells into the contused spinal cord of nude rats. J Neurosurg Spine. 2008 Feb;8(2):153-62. doi: 10.3171/SPI/2008/8/2/153. PMID 18248287
- [Background] Zurita M, Vaquero J. Bone marrow stromal cells can achieve cure of chronic paraplegic rats: functional and morphological outcome one year after transplantation. Neurosci Lett. 2006 Jul 10;402(1-2):51-6. doi: 10.1016/j.neulet.2006.03.069. Epub 2006 May 19. PMID 16713677
- [Background] Yoon SH, Shim YS, Park YH, Chung JK, Nam JH, Kim MO, Park HC, Park SR, Min BH, Kim EY, Choi BH, Park H, Ha Y. Complete spinal cord injury treatment using autologous bone marrow cell transplantation and bone marrow stimulation with granulocyte macrophage-colony stimulating factor: Phase I/II clinical trial. Stem Cells. 2007 Aug;25(8):2066-73. doi: 10.1634/stemcells.2006-0807. Epub 2007 Apr 26. PMID 17464087
- [Background] Osaka M, Honmou O, Murakami T, Nonaka T, Houkin K, Hamada H, Kocsis JD. Intravenous administration of mesenchymal stem cells derived from bone marrow after contusive spinal cord injury improves functional outcome. Brain Res. 2010 Jul 9;1343:226-35. doi: 10.1016/j.brainres.2010.05.011. Epub 2010 May 12. PMID 20470759
- [Background] Hu SL, Luo HS, Li JT, Xia YZ, Li L, Zhang LJ, Meng H, Cui GY, Chen Z, Wu N, Lin JK, Zhu G, Feng H. Functional recovery in acute traumatic spinal cord injury after transplantation of human umbilical cord mesenchymal stem cells. Crit Care Med. 2010 Nov;38(11):2181-9. doi: 10.1097/CCM.0b013e3181f17c0e. PMID 20711072
- [Background] Parr AM, Tator CH, Keating A. Bone marrow-derived mesenchymal stromal cells for the repair of central nervous system injury. Bone Marrow Transplant. 2007 Oct;40(7):609-19. doi: 10.1038/sj.bmt.1705757. Epub 2007 Jul 2. PMID 17603514